CLINICAL TRIAL: NCT03247348
Title: Reducing Sedentary Time in Fibromyalgia (ReSeT-FM): A Feasibility Study
Brief Title: Reducing Sedentary Time in Fibromyalgia Patients
Acronym: ReSeT-FM
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Richard L. Roudebush VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kelly M Naugle, PhD, Assistant Professor, Indiana University
Other Study IDs: 1702201230
Record Dates: First submitted 2017-08-01; First posted 2017-08-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia; Veterans
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ReSeT-FM intervention — The ReSeT-FM intervention focuses on behavior changes strategies aimed at reducing sedentary time and includes: education, goal setting, self-monitoring of behavior and behavioral prompts to move via an activity tracker and phone app, and feedback on behavior via weekly meetings with study coaches.

SUMMARY:
This study evaluates the feasibility of a behavioral intervention designed to replace sedentary behavior with light physical activity in veterans with Fibromyalgia. The study will also evaluate the acceptability of the intervention among veterans and intervention effects on pain and physical function.

DETAILED DESCRIPTION:
Recent research suggests that individuals with Fibromyalgia (FM) who spend more time in sedentary behavior and less time in light physical activity experience greater clinical pain and overall impact of FM, irrespective of time spent in moderate to vigorous physical activity. To date, no studies have investigated the potential impact of reducing sedentary behavior on key clinical and physical function outcomes in FM. The overall objective of the pilot project is to design and evaluate the feasibility of an 8-week behavioral intervention designed to replace sedentary behavior with light physical activity in veterans with FM. Mixed (quantitative and qualitative) methods will be used to evaluate the behavioral intervention, which is based on constructs from social cognitive and self-regulatory theories that consistently identify important drivers of behavior change as: education, goal-setting, self-monitoring and behavioral prompts to move via an activity tracker and phone app, and feedback on behavior via weekly meetings.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible if they have:

* 2010 American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia: Widespread Pain Index (WPI) greater than 7 and Symptom Severity Scale (SS) greater than 5 or WPI 3-6 and SS greater than 9.
* Symptoms have been present at a similar level for at least 3 months
* The subject does not have a disorder that would otherwise explain the pain
* Moderate pain severity (pain severity score greater than 5)
* No changes in fibromyalgia medications for last 4 weeks
* Self-reporting at least 8 hours per day sitting on 5 or more days per week
* Having access to either an Android or iPhone smart phone with access to internet

Exclusion Criteria:

* Significant cardiovascular disease
* chronic obstructive pulmonary disease (COPD) or asthma needing home oxygen
* Stroke or transient ischemic attack (TIA) in last 6 months
* Cancer (other than skin cancer) and receiving treatment for it
* Active psychosis
* Active suicidal ideation
* Moderate to severe cognitive impairment
* Engaging in more than 30 minutes of moderate to vigorous physical activity 3 or more days per week
* Currently using an app or activity tracker to track physical activity
* Enrolled in another research study related to pain or exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change in minutes of sedentary time per day | This measure will be assessed at baseline and 8 weeks. At each time point the accelerometer will be worn for 1 week.
  Participants will wear an Actigraph accelerometer, which provides a well established measure of sedentary time.
Change in minutes of light physical activity per day. | This measure will be assessed at baseline and 8 weeks. At each time point the accelerometer will be worn for 1 week.
  Participants will wear an Actigraph accelerometer, which provides a well established measure of light physical activity.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised (FIQ-R) | This measure will be assessed at baseline and 8 weeks.
  This 21-item instrument assesses symptoms, function, and overall impact of fibromyalgia.
Brief Pain Inventory (BPI) | This measure will be assessed at baseline and 8 weeks.
  This 11-item instrument rates the intensity of pain as well as interference of pain with mood, physical activity, work, social activity, relations with others, sleep, and enjoyment of life.
Medical Outcomes Study Short Form Questionnaire (SF-12) | This measure will be assessed at baseline and 8 weeks.
  This questionnaire assess physical and mental functioning.
Six minute walk test | This measure will be assessed at baseline and 8 weeks.
  This physical function test measures functional aerobic capacity. Subjects will walk as far as possible at their usual pace in 6 minutes around a predetermined indoor walking course on a flat surface.
30-second Chair stand test | This measure will be assessed at baseline and 8 weeks.
  This physical function test measures lower body muscle strength. Subjects will complete as many sit to stands in a chair as possible in 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Naugle, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Roudebush VA Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No